CLINICAL TRIAL: NCT00857142
Title: A Study to Evaluate the Relative Bioavaility of Oxymorphone Hydrochloride 40 mg Extended-Release Tablets(Sandoz, Inc. Compared to Opana ER (Oxymorphone Hydrochloride) Extended-Release Tablets, 40 mg (Edo Pharmaceuticals Inc.) in Healthy Volunteers Under Non-fasted COnditions
Brief Title: Bioavailability of Oxymorphone Hydrochloride 40 mg Extended Release Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, VP Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10713410
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxymorphone

ARMS (2):
- 1 (Experimental): Oxymorphone hydrochloride 40 mg extended release tablets (Sandoz)
  Interventions: Drug: oxymorphone hydrochloride
- 2 (Active Comparator): Opana 40 mg extended release tablets
  Interventions: Drug: Opana

INTERVENTIONS:
Drug: oxymorphone hydrochloride
  Arms: 1
Drug: Opana
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioequivalence of oxymorphone hydrochloride extended release tablets (Sandoz) with Opana extended release oxymorphone hydrochloride tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, nonmedical history or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C
* Treatment for drug or alcohol abuse
* Allergy to opiates

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daryl G. Ficklin, D.O., Principal Investigator — Novum Pharmaceutical Research Services